CLINICAL TRIAL: NCT01031849
Title: Análisis de Los Cambios en el Tejido Adiposo de Pacientes Con infección VIH y Lipoatrofia en Tratamiento Con análogos de nucleósidos timidínicos, Tras el Cambio a Monoterapia Con Lopinavir/Ritonavir
Brief Title: Analysis of Changes in Adipose Tissue of Patients With Lipoatrophy HIV Infection Treated With Nucleoside Thymidine, After Switching to Monotherapy With Lopinavir / Ritonavir
Acronym: BIOKAL
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: patient sample not reached
Sponsor: Ines Perez (Other)
Responsible Party: Sponsor-Investigator, Ines Perez, MD, Hospital San Carlos, Madrid
Organization: Hospital San Carlos, Madrid (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HCSKAL-2009-01; 2009-016090-14 (Other: EudraCT Number)
Record Dates: First submitted 2009-12-04; First posted 2009-12-15 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: HIV Infections
Keywords: HIV 1 patients
MeSH Terms: conditions — HIV Infections | interventions — lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Kaletra, all patients (Experimental): Patients will change actual treament for monotherapy LPV/r. They only will take Kaletra 2/day
  Interventions: Drug: Kaletra

INTERVENTIONS:
Drug: Kaletra — Each tablet of Kaletra contains 200 mg of Lopinavir and 50mg of ritonavir. The patients will take two tablets of Kaletra bid.

SUMMARY:
The objective is to analyse the changes in the adipose tissue hystological features and the adipogenesis gene expression and related to inflammation after 48 and 96 weeks after the change from AZT+3TC+ABC (Trizivir®) to a monotherapy treatment with LPV/r (Kaletra®)

ELIGIBILITY:
Inclusion Criteria:

* Patients infected with VIH-1, documented with a positive HIV-1 antibody test and/or positive PCR, confirmed for HIV-1 RNA.
* Patients treated with a HAART that should contain AZT+3TC+ABC (Trizivir®)
* Patients with an indetectable viral load, which will be defined <40 copies/mL within the last six months.
* Patients with a lipoatrophy clinical evidence (which will be defined as moderate or severe, according to the Lipodystrophy Severity Grading Scale).
* Men or women aged ≥ 18.
* For women of childbearing potential, negative urine pregnancy test during the Screening visit.
* Patients that have signed and dated the Informed consent Form prior to any Study-specific procedure.

Exclusion Criteria:

* Patients with evidence of protease inhibitors failure, and/or documented evidence of protease gene resistance mutation. This evidence could be prior or during the inclusion period in the Study.
* Patients who, for any reason could not be treated with LPV/r.
* Cachexia, defined as an Body Mass Index <17 Kg/m2.
* Pregnant or breastfeeding women, or women of childbearing potential who do not use the appropriate contraceptive method, according to the Investigator judgment.
* Clinically relevant disease or condition, according to the Investigator judgment, three months prior to the patient inclusion in the Study.
* Patients taking the following concomitant medication that could affect the adipocyte function or morphology, such as: insulin, steroids, anabolic steroid, anti-inflammatory medication for more than three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-02; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change in those representative gene expression of adipose tissue toxicity (variable established from those gene involved in adipogenesis, inflammation and metabolism. This gene expression will counted) | 48 and 96 weeks

SECONDARY OUTCOMES:
Changes in physical fat deposits | Baseline, 24, 48, 72 and 96 weeks
Changes in leptine and adiponectine plasma levels | baseline, 24, 48, 72 and 96 weeks
Patients percentage with virologic response (ARN-VIH< 50 copies/mL) | 48 and 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Estrada, MD, Principal Investigator — hospital Clínico San Carlos, Madrid
Locations (2):
- Spain (2):
  - Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid